CLINICAL TRIAL: NCT00948506
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Single-center Proof of Concept Study of Topical Cidofovir for the Prevention of Hair Growth
Brief Title: Trial of Topical Cidofovir for the Prevention of Hair Growth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 809821
Record Dates: First submitted 2009-07-23; First posted 2009-07-29 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Prevention of Hair Growth
MeSH Terms: interventions — Cidofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1% topical cidofovir (Placebo Comparator): 1% topical cidofovir to one side of the face and placebo to the other side of the face
  Interventions: Drug: 1% topical cidofovir; Drug: Placebo
- 3% topical cidofovir (Placebo Comparator): 3% topical cidofovir to one side of the face and placebo to the other side of the face
  Interventions: Drug: 3% topical cidofovir; Drug: Placebo

INTERVENTIONS:
Drug: 1% topical cidofovir — 1% topical cidofovir
  Other Names: Vistide
  Arms: 1% topical cidofovir
Drug: 3% topical cidofovir — 3% topical cidofovir
  Other Names: Vistide
  Arms: 3% topical cidofovir
Drug: Placebo — topical placebo

SUMMARY:
This is a two-arm, single center placebo-controlled double-blind proof of concept study which will evaluate the safety and efficacy of topical cidofovir (both 1% and 3%)compared to placebo for the prevention of hair growth.

DETAILED DESCRIPTION:
This is a phase II randomized, placebo controlled double blind, dose-ranging clinical trial of topical cidofovir for the prevention of hair growth. This proof of concept study will evaluate 1% and 3% cidofovir in petrolatum topically applied once a day to the target treatment area on the hair bearing area of the face known as the beard area. This target area will be of a circular shape with a diameter of three centimeters along the jaw line of one side of the face.The first 14 enrolled subjects in the study will be randomized in a 1:1 fashion to receive either 1% topical cidofovir and placebo or 3% topical cidofovir and placebo. The last cohort of subjects to be enrolled in the study to achieve a total of 16 evaluable subjects will all receive the 3% formulation and placebo. Subjects will also be randomized as to which side of their face (left or right) will receive active drug versus placebo.

Subjects will be treated for up to eight weeks. Any subject who achieves 100% alopecia (which corresponds to a 0 on the PGA of Hair Density) in the treated area prior to eight weeks will be classified as a responder and will discontinue active treatment and begin the four week observation period. From the time of discontinuing treatment, subjects will be followed for four weeks during which time safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to give informed consent.
2. Subjects must be male, age 18 years or older.
3. Score of 4 or 5 on the Physician's Global Assessment of Hair Density at baseline
4. Subjects must have to shave at least once a day to avoid a visible beard with a hair length that is above the skin line.
5. Male subjects who are sexually active with female partners and are capable of fertilization must ensure that their female partners will either be postmenopausal, surgically incapable of childbearing, or will use a medically acceptable method of contraception throughout the entire study period. Medically acceptable methods of contraception that may be used by the subject and/or partner include oral contraceptives or patch, diaphragms with spermicide, IUD, condom with spermicide, or progestin implant or injection. Female partners taking oral contraceptives must have taken them consistently for at least two months prior to subject receiving study medication.
6. Subjects must be able to limit the use of alcohol to 2 or fewer drinks per day for the duration of the study period. One drink corresponds to 6 oz of wine, 12 oz of beer or 1 oz of hard liquor.
7. Subjects must be willing and able to avoid exposure of the study drug to others
8. Subjects must be able to understand and comply with drug storage and application procedures

Exclusion Criteria:

1. Use of an investigational medication 180 days prior to study enrollment (day 0).
2. Use of topical medication that can affect hair growth during the 8 weeks prior to the baseline visit (e.g. minoxidil, eflornithine HCl).
3. Use of a systemic medication that can affect hair growth during the 180 days prior to the baseline visit (e.g. minoxidil, cyclosporine A, finasteride).
4. Clinically significant abnormality in liver function, renal function, chemistry panel or CBC (AST or ALT ≥ 2 times the laboratory's upper limit of normal, hemoglobin < 10.0 g/dL, platelet count <125,000/cm3, white blood count <3,500 cells/cm3 or > 15,000 cells/cm3, or serum creatinine ≥ 1.5 mg/dL) within two weeks of the baseline visit.
5. Proteinuria or hematuria upon urine analysis within two weeks of the baseline visit.
6. Active inflammatory skin disease in the treatment area (e.g. acne, cysts) or neoplasms in the treatment area that in the judgment of the investigator precludes enrollment.
7. History of skin cancer or actinic keratoses in the treatment area.
8. Concomitant use of any topical medication in the target areas during the study.
9. Previous history of alopecia areata.
10. Use of a nephrotoxic medication (tobramycin, gentamycin, amikacin, amphotericin B, foscarnet, vancomycin, non-steroidal anti-inflammatory agents) 7 days prior to the baseline visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Gelfand, MD, MSCE, Principal Investigator — Hospital of the University of PA
Locations (1):
- Hospital of the University of PA, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1% Cidofovir and Placebo: Subjects received 1% topical cidofovir to one side of the face and placebo to the other side of the face in a split-face design.
- 3% Cidofovir and Placebo: Subjects received 3% topical cidofovir to one side of the face and placebo to the other side of the face in a split-face design.
Period: Overall Study
Arm/Group | 1% Cidofovir and Placebo | 3% Cidofovir and Placebo
Started | 11 | 9
Completed | 8 | 8
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Cidofovir and Placebo | 3% Cidofovir and Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.55 (8.32) | 31.44 (12.02) | 34.25 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Physician's Global Assessment (PGA) of Hair Density
Description: Number of participants with a score of 2 or less on the Physician Global Assessment (PGA) of Hair Density at the end of active treatment. The five point scale ranges from 0 (total alopecia) to 5 (very dense).
Time Frame: up to 8 weeks or end of active treatment
Population: The analysis was performed using intention-to-treat and all enrolled participants who received treatment were included in the analysis. For participants who withdrew during treatment, the data from their last visit were carried forward.
Measure: Number; unit: participants
Groups:
- 1% Cidofovir: Subjects received 1% topical cidofovir to one side of the face in a split-face design (placebo was applied to the other side of the face).
- 3% Cidofovir: Subjects received 3% topical cidofovir to one side of the face in a split-face design (placebo was applied to the other side of the face).
- Placebo: Subjects received placebo to one side of the face in a split-face design (1% or 3% cidofovir was applied to the other side of the face).
Arm/Group | 1% Cidofovir | 3% Cidofovir | Placebo
Number analyzed (Participants) | 11 | 9 | 20
participants | 1 | 0 | 1

2. Secondary Outcome: Subject-reported Adverse Events or Abnormal Findings
Description: Number of participants who reported an adverse event (as assessed by subject interview and if indicated, physical exam) or had abnormal finding on urine and blood laboratory examination
Time Frame: up to 16 weeks
Population: The analysis was performed using intention-to-treat, whereby all enrolled participants who received treatment were analyzed.
Measure: Number; unit: participants
Groups:
- 1% Cidofovir and Placebo: Subjects received 1% topical cidofovir to one side of the face in a split-face design (placebo was applied to the other side of the face).
- 3% Cidofovir and Placebo: Subjects received 3% topical cidofovir to one side of the face in a split-face design (placebo was applied to the other side of the face).
Arm/Group | 1% Cidofovir and Placebo | 3% Cidofovir and Placebo
Number analyzed (Participants) | 11 | 9
participants | 6 | 6

ADVERSE EVENTS:
Arm/Group | 1% Cidofovir and Placebo | 3% Cidofovir and Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/9
Other Adverse Events (participants affected / at risk) | 6/11 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% Cidofovir and Placebo (N=11) | 3% Cidofovir and Placebo (N=9)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant self-reported an episode of gastrointestinal bleeding resulting in hospitalization but no documentation of the hospitalization was received. The IRB was notified.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% Cidofovir and Placebo (N=11) | 3% Cidofovir and Placebo (N=9)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Erythema of the treatment area (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Erythema - in 1 subject on the 3% cidofovir-treated side; in 2 subjects on the 1% cidofovir-treated side
Pruritis of treatment area (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Pruritis - in 1 subject on the 3% cidofovir-treated side; in 1 subject on both the 1% cidofovir-treated and placebo-treated sides
Cold sores (Infections and infestations) | 1 (1) | 1 (1)
Rash over the untreated area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin tenderness of untreated area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eyelid twitch (Nervous system disorders) | 0 (0) | 1 (1)
Flare of pre-existing brachial neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Dog bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toothache after a dental procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Neck swelling after surgical nerve block (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No